CLINICAL TRIAL: NCT07197164
Title: Safety and Efficacy of 10-day Course of Remdesivir to Prevent Severe COVID-19 in Asymptomatic or Paucisymptomatic SARS-COV-2-positive Kidney Transplant Recipients: a Single-arm Proof-of-concept Interventional Trial
Brief Title: Safety and Effectiveness of a Remdesivir Treatment to Prevent Severe COVID-19 in Kidney Transplant Patients
Acronym: COVIDKIDNEY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVIDKIDNEY; 2024-519272-96-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-25; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: COVID - 19; Renal Transplant; SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Intervention Model Description: Phase 2, proof of concept open-label, single-center, single- arm clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Single Arm with remdesivir
  Interventions: Drug: Remdesivir (RDV)

INTERVENTIONS:
Drug: Remdesivir (RDV) — Participants will receive their first dose of remdesivir also within the 24 (+/-12) hours prior to going to the operating room. Remdesivir doses will be 200 mg on day 1, followed by 100 mg daily from days 2 to 10, for a total of 10 days.
  Other Names: Veklury

SUMMARY:
Since the start of the COVID-19 pandemic, the approach to solid organ transplantation has evolved. Transplants using organs (excluding lungs) from COVID-19-positive donors have shown short-term safety, but there is limited data on recipients who are SARS-CoV-2 positive. Currently, kidney transplants in such recipients are delayed until symptoms resolve and a negative PCR is preferred, despite the risks of prolonged dialysis and increased cold ischemia time.

Recent data from the Omicron era suggest that early antiviral treatment may reduce complications. Immunosuppressive therapy might even help mitigate severe inflammatory responses. The proposed study aims to show that kidney transplantation can be safely performed in asymptomatic or mildly symptomatic COVID-19-positive recipients who begin antiviral treatment (remdesivir) within 24 hours before transplant and continue for 10 days. This could reduce waiting times and improve outcomes.

Remdesivir is an antiviral safe for use in patients with low kidney function, including those on dialysis or post-transplant, with minimal side effects. The hypothesis is that this treatment strategy can prevent progression to severe COVID-19 and allow safe transplantation

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years-old
2. Patients with end-stage kidney disease that are included on the local kidney transplant waiting list who get an offer of a compatible organ and, subsequently, have a transplant procedure scheduled in the next 24 (+/-) 12 hours, or patients with end-stage kidney disease that are planned to receive a non-cadaveric donor kidney transplant on the following 5 days.
3. Have a positive SARS-CoV-2 nasopharyngeal PCR or RAT within 5 days prior to transplant surgery.
4. Have previously received at least three SARS-CoV-2 vaccine doses, with a minimum time elapsed of 3 months since the last dose received.
5. Are asymptomatic or have mild acute COVID-19 symptoms during the previous 5 days (headache, sore throat, cough, chest pain, nausea, diarrhea, fatigue, loss of smell or taste, myalgia) excluding fever in the previous 48 hours (>38ºC) or shortness of breath.
6. Post-menopausal or fertile females (females who are not surgically sterile or postmenopausal defined as amenorrhea for >12 months) that agree to avoid pregnancy during the study. If sexually active fe-male; using highly effective contraceptive methods (hormonal contraception, intra-uterine device (IUD), or anatomical sterility in self or partner*) while on study treatment. All female volunteers must be willing to undergo urine pregnancy tests at time of enrollment.
7. Having understood the information provided and capable of giving consent to participate in this trial by signing the Informed Consent document.

Exclusion Criteria:

1. Pregnant or breastfeeding women, at time of enrollment
2. Patients requiring supplementary oxygen at baseline or diagnosed with severe COPD or pulmonary fibrosis.
3. Patients having any of the following at the screening period: i) O2 saturation below 94% on room air; ii) respiratory frequency of > 30bpm; or iii) Xray showing new-onset pulmonary infiltrates suggesting COVID-19 pneumonia.
4. Patients having fever (>38ºC) in the last 48 hours or shortness of breath in the previous 5 days.
5. Previous history of hypersensitivity, documented allergy or contraindications to receive remdesivir.
6. ABO incompatible kidney transplant
7. Desensitization therapy indicated as induction therapy for high immunological risk transplant with Donor Specific HLA Antibodies (DSA)
8. Participants who receive different types of induction immunosuppression other than the standard induction protocols with lymphocyte- depleting agents (thymoglobulin or basiliximab).
9. Active liver disease with AST or ALT >3 ULN, Total bilirubin ≥2 × ULN (for Gilbert's syndrome, direct bilirubin >ULN is exclusionary) within the past 3 months, or liver function impairment with Class B or C per Child Pugh classification.
10. Suspected or confirmed concurrent active respiratory infection other than COVID-19 that may interfere with the evaluation of response to the study intervention.
11. Any comorbidity requiring hospitalization and/or surgery within 7 days prior to study entry, or that is considered life threatening within 30 days prior to study entry, as determined by the investigator.
12. Prior participation in this trial.
13. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of participants who develop severe COVID-19 following kidney transplantation | to 28 days and 90 days post-transplant
  Primary estimates: Severe SARS-CoV-2 will be defined as: Hypoxemia (O2 sat <94%), one or more compatible respiratory symptoms (fever, dyspnea, increased respiratory frequency > 22, cough) AND new radiologic infiltrates compatible with COVID-19 in a chest X Ray, chest CT or ultrasound.

SECONDARY OUTCOMES:
Number of deaths (all causes mortality) at days 28 and 90 post-transplant | at days 28 and 90 after transplant
  the cumulative mortality at days 28 and 90 after transplant in asymptomatic or paucisymptomatic SARS-CoV-2-positive kidney transplant recipients receiving a 10-day course of remdesivir
Time (days) to resolution and to recovery of all targeted symptoms through Day 28 and Day 90 | At day 28 and day 90
  Duration of targeted COVID-19 symptoms (COVID-19 Questionnaire).
Proportion of participants requiring extension of the hospitalization beyond POD10 (all cause and related to COVID-19) | At day 28
  % participants with COVID complications at the hospitalization that requires invasive Mechanical ventilation, intensive care unit (ICU) stayed or extension of the hospitalization related to COVID-19
Proportion of participants with symptomatic rebound through day 28. | At day 28
  % participant who, after an initial improvement or resolution of symptoms, experience a recurrence of symptoms within the 28-day follow-up period
To describe the clearance kinetics of SARS-CoV-2 infection in the post-transplant period | At day 0, 5, 10, 14, 21 and 28
  Number and proportion of participants with negative nasopharyngeal SARS-CoV-2 PCR, and median CT values if positive, at POD 0 (time of diagnosis), POD5, POD10, POD14, POD21, and POD28 and Whole genome sequencing of SARS-CoV-2 to evaluate emergence of substitutions associated with resistance to remdesivir in participants who have a positive SARS-CoV-2 PCR and CT values below or equal to 25.
Number of Participants with Treatment-Related Adverse Events | From enrollment to the end of study at 6 months
  Incidence of SAEs and AEs leading to drug discontinuation and number and proportion of any treatment-emergent hepatic AE (Elevation of any grade in ALT or AST levels, prothrombin time or INR, or blood bilirubin), number and proportion of severe liver failures (defined as elevated LFTs and presence of coagulopathy or hepatic encephalopathy) and mumber of patients that develop hypersensitivity or infusion-related reactions
incidence of graft complications | at day 7, day 28 and day 90
  Number and proportion of participants with stage 2 or 3 AKI and or that present a proven-biopsy showing acute humoral or cellular rejection and or dialysis needed

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain